CLINICAL TRIAL: NCT06635863
Title: Immunosuppression Versus Medical Therapy for UN-explained Low Ejection Fraction and VT
Brief Title: Comparing Immune System Suppression to Medication for Unexplained Heart Function and Irregular Heartbeat
Acronym: IMMUNE VT
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Roderick Tung (Other)
Responsible Party: Sponsor-Investigator, Roderick Tung, Professor of Medicine; Chief, Division of Cardiology, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003729
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Ventricular Arrythmia; Non-ischemic Cardiomyopathy; Arrhythmogenic Inflammatory Cardiomyopathy
Keywords: immunosuppressive therapy; immunomodulatory; inflammation by FDG; guideline-direct medical therapy
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppression (Experimental): Prednisone 40mg x 8weeks + GDMT
  Interventions: Drug: Prednisone 40mg
- Standard of Care (No Intervention): GDMT alone

INTERVENTIONS:
Drug: Prednisone 40mg — Prednisone 40mg x 8weeks
  Arms: Immunosuppression

SUMMARY:
Ventricular tachycardia (VT, a potentially fatal condition where the ventricle of the heart beats rapidly) superimposed on non-ischemic cardiomyopathy (NICM, a disease of heart with broad etiologies except coronary artery disease). This disease has been associated with inflammation in the heart.

The purpose of this study is to assess the benefit of immunosuppressive therapy to suppress the VT, improve heart function, avoid invasive intervention and hospitalization. Positron Emission Tomography (PET) imaging shows inflammation in the heart. After enrollment, baseline tests (including physical exams, blood tests, genetic test, electrocardiography, echocardiography) will be done. Next, will be an 8-week medication regimen which contains either immunosuppressive drugs or standard GDMT without immunosuppressant medication. Some of the examinations will be repeated during the study to evaluate the treatment response and monitor any adverse events.

DETAILED DESCRIPTION:
Ventricular arrhythmia (VT) is a well-established consequence in patients with non-ischemic cardiomyopathy (NICM). NICM is a broad category that includes a wide spectrum of causes, which may include: bacterial, viral toxin mediated and immune mediated and "unexplained" when coronary disease has been excluded. The pathophysiology of NICM is not well understood but inflammatory responses with macrophage recruitment during remodeling have been described. On the other hand, an infectious trigger i.e. myocarditis may be the inciting event for the development of cardiomyopathy. A previous study by Tung et al showed that nearly 50% of patients with unexplained cardiomyopathy and ventricular arrhythmias presented ongoing focal myocardial inflammation on PET. To date, targeting inflammation as a substrate in order to reduce burden of ventricular tachycardia has not been investigated in randomized prospective fashion.

The TIMIC trial was one of the few randomized studies to examine long-term benefit of immunosuppressive therapies in patients with virus-negative NICM. A moderate improvement in Left Ventricular Ejection Fraction (LVEF) over 6 months after initiation of immunosuppressive therapy was demonstrated in this study but current guidelines do not routinely recommend anti-inflammatory therapies for NICM. While considered to be gold standard, endomyocardial biopsy can often times be incorrect due to sampling error and typically is not performed multiple times in patient with chronic non-ischemic cardiomyopathy. Fasting Fluorodeoxyglucose (FDG)-positron emission tomography (PET) is an emerging imaging modality to identify and monitor abnormal metabolic patterns of the myocardium. By exploiting the metabolic demand of inflammatory tissue with macrophage recruitment, PET imaging is emerging as the preferred modality to diagnose and measure response to therapy for patients with myocarditis and sarcoidosis. A recent study by Kandolin et al in Finland showed that the incidence of cardiac sarcoidosis has increased by 20-fold over the past two decades.

FDG-PET may reveal inflammation as a central pathophysiologic mechanism in a significant proportion of patients with unexplained cardiomyopathy and VT. Potential innovative insights from the trial will be to identify the underlying pathogenesis of idiopathic cardiomyopathy and assess whether immunosuppression changes the clinical course of patients with identified arrhythmogenic cardiomyopathy. Aside from guideline-direct medical therapy (GDMT), antiarrhythmic agents, and catheter ablation, there are no disease-specific therapies for patients with VT and NICM. Prospective studies that evaluate the incidence of occult inflammation and clinical response to anti-inflammatory and immunosuppressive therapy have not been performed to date and are warranted for the emerging NICM population referred for advanced heart failure and arrhythmia management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, all races, all gender
* LV systolic function < 50%
* Optimized GDMT Per physicians' discretion (SOC treatment)
* No evidence of ischemic cardiomyopathy
* No evidence of obstructive coronary disease
* Viral panel negative
* NYHA class II, III and ambulatory class IV heart failure
* History of VA (documentation of Sustained VT last more than 30 seconds)
* Heart inflammation confirmed by PET scan
* Steroid use within 12 months prior to of date of consent

Exclusion Criteria:

* Life expectancy less than 24 months
* Pregnancy
* Contra indications or intolerance of prednisone or any excipients in the formulation
* Hypothalamic-pituitary-adrenal axis suppression, Cushing's syndrome, active infection, glaucoma or any other pathology where corticosteroids are not recommended.
* Any patient with HIV, low white blood cells, and chronic infection (active fungal, TB, Valley fever)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Burden of ventricular arrhythmias | 12 months (8 weeks and 6 months)
  Documented sustained monomorphic ventricular tachycardia >30 seconds or any appropriate defibrillator therapy (shock or antitachycardia pacing).
Change in left ventricular ejection fraction (LVEF) | 12 months (8 weeks and 6 months)
  Left ventricular ejection fraction measured with Simpson method with echocardiography.
Change in QRS duration | 12 months (8 weeks and 6 months)
  QRS duration (milliseconds) measured with a 12-lead ECG.
Change in FDG (18F-fluorodeoxyglucose) uptake | 12 months
  Change in FDG uptake compared to initial uptake assessed with 18F-fluorodeoxyglucose PET (FDG-PET). Myocardial FDG uptake will be reported as non, focal or diffuse and/or isolated with focal pattern.

SECONDARY OUTCOMES:
Cardiovascular hospitalization | 6 months and 12 months.
  Patient hospitalization (yes/no) due to a cardiovascular reason. Cardiovascular hospitalization is defined as a hospital admission after the randomized procedure for heart failure, treatment associated complication, or arrhythmia-related causes during the follow-up period.
Need for catheter ablation | 6 months and 12 months.
  Need for catheter ablation (yes/no) due to ventricular arrhythmias.
NYHA functional class | 6 months and 12 months
  New York Heart Association functional class I, II, III or IV.
Survival | 6 months and 12 months
  Freedom from all-cause mortality and cardiac transplant.

OTHER OUTCOMES:
Medication adverse events | 6 months and 12 months
  Medication related adverse events: steroid-induced diabetes, infection, weight gain, osteopenia, or psychosis.
System related adverse events | 6 months and 12 months.
  System related adverse events: worsening LVEF, high frequency of ventricular tachycardia seen on monitoring, or hospitalizations related to either.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be stored within REDCap, for use by other researchers including those outside of the study, but only within the University of Arizona. The consent for the study includes information that de-identified data may be used for future unspecified research.
Time Frame: After completion of study and stored for future unspecified research. Only de-identified data will be made available.
Access Criteria: A request for access to the de-identified data will be made and access will only be granted to those with permission from the PI.

REFERENCES:
- [Background] Tung R, Bauer B, Schelbert H, Lynch JP 3rd, Auerbach M, Gupta P, Schiepers C, Chan S, Ferris J, Barrio M, Ajijola O, Bradfield J, Shivkumar K. Incidence of abnormal positron emission tomography in patients with unexplained cardiomyopathy and ventricular arrhythmias: The potential role of occult inflammation in arrhythmogenesis. Heart Rhythm. 2015 Dec;12(12):2488-98. doi: 10.1016/j.hrthm.2015.08.014. Epub 2015 Aug 10. PMID 26272522
- [Background] Belperio JA, Shaikh F, Abtin FG, Fishbein MC, Weigt SS, Saggar R, Lynch JP 3rd. Diagnosis and Treatment of Pulmonary Sarcoidosis: A Review. JAMA. 2022 Mar 1;327(9):856-867. doi: 10.1001/jama.2022.1570. PMID 35230389
- [Background] Rahaghi FF, Baughman RP, Saketkoo LA, Sweiss NJ, Barney JB, Birring SS, Costabel U, Crouser ED, Drent M, Gerke AK, Grutters JC, Hamzeh NY, Huizar I, Ennis James W 4th, Kalra S, Kullberg S, Li H, Lower EE, Maier LA, Mirsaeidi M, Muller-Quernheim J, Carmona Porquera EM, Samavati L, Valeyre D, Scholand MB. Delphi consensus recommendations for a treatment algorithm in pulmonary sarcoidosis. Eur Respir Rev. 2020 Mar 20;29(155):190146. doi: 10.1183/16000617.0146-2019. Print 2020 Mar 31. PMID 32198218
- [Background] Melani AS, Bigliazzi C, Cimmino FA, Bergantini L, Bargagli E. A Comprehensive Review of Sarcoidosis Treatment for Pulmonologists. Pulm Ther. 2021 Dec;7(2):325-344. doi: 10.1007/s41030-021-00160-x. Epub 2021 Jun 18. PMID 34143362
- [Background] Kandolin R, Lehtonen J, Airaksinen J, Vihinen T, Miettinen H, Ylitalo K, Kaikkonen K, Tuohinen S, Haataja P, Kerola T, Kokkonen J, Pelkonen M, Pietila-Effati P, Utrianen S, Kupari M. Cardiac sarcoidosis: epidemiology, characteristics, and outcome over 25 years in a nationwide study. Circulation. 2015 Feb 17;131(7):624-32. doi: 10.1161/CIRCULATIONAHA.114.011522. Epub 2014 Dec 19. PMID 25527698
- [Background] Ishimaru S, Tsujino I, Takei T, Tsukamoto E, Sakaue S, Kamigaki M, Ito N, Ohira H, Ikeda D, Tamaki N, Nishimura M. Focal uptake on 18F-fluoro-2-deoxyglucose positron emission tomography images indicates cardiac involvement of sarcoidosis. Eur Heart J. 2005 Aug;26(15):1538-43. doi: 10.1093/eurheartj/ehi180. Epub 2005 Apr 4. PMID 15809286
- [Background] Chareonthaitawee P, Beanlands RS, Chen W, Dorbala S, Miller EJ, Murthy VL, Birnie DH, Chen ES, Cooper LT, Tung RH, White ES, Borges-Neto S, Di Carli MF, Gropler RJ, Ruddy TD, Schindler TH, Blankstein R; EXPERT CONTENT REVIEWERS. Joint SNMMI-ASNC Expert Consensus Document on the Role of 18F-FDG PET/CT in Cardiac Sarcoid Detection and Therapy Monitoring. J Nucl Med. 2017 Aug;58(8):1341-1353. doi: 10.2967/jnumed.117.196287. No abstract available. PMID 28765228
- [Background] Kebed KY, Carter SV, Flatley E, Ward RP, Moss JD, Appelbaum DE, Singh A, Lang RM, Tung R, Patel AR. Prevalence of newly diagnosed sarcoidosis in patients with ventricular arrhythmias: a cardiac magnetic resonance and 18F-FDG cardiac PET study. Int J Cardiovasc Imaging. 2021 Apr;37(4):1361-1369. doi: 10.1007/s10554-020-02090-2. Epub 2020 Nov 22. PMID 33225427
- [Background] Youssef G, Leung E, Mylonas I, Nery P, Williams K, Wisenberg G, Gulenchyn KY, Dekemp RA, Dasilva J, Birnie D, Wells GA, Beanlands RS. The use of 18F-FDG PET in the diagnosis of cardiac sarcoidosis: a systematic review and metaanalysis including the Ontario experience. J Nucl Med. 2012 Feb;53(2):241-8. doi: 10.2967/jnumed.111.090662. Epub 2012 Jan 6. PMID 22228794
- [Background] Wicks EC, Menezes LJ, Barnes A, Mohiddin SA, Sekhri N, Porter JC, Booth HL, Garrett E, Patel RS, Pavlou M, Groves AM, Elliott PM. Diagnostic accuracy and prognostic value of simultaneous hybrid 18F-fluorodeoxyglucose positron emission tomography/magnetic resonance imaging in cardiac sarcoidosis. Eur Heart J Cardiovasc Imaging. 2018 Jul 1;19(7):757-767. doi: 10.1093/ehjci/jex340. PMID 29319785
- [Background] Palmisano A, Vignale D, Peretto G, Busnardo E, Calcagno C, Campochiaro C, De Luca G, Sala S, Ferro P, Basso C, Del Maschio A, De Cobelli F, Esposito A. Hybrid FDG-PET/MR or FDG-PET/CT to Detect Disease Activity in Patients With Persisting Arrhythmias After Myocarditis. JACC Cardiovasc Imaging. 2021 Jan;14(1):288-292. doi: 10.1016/j.jcmg.2020.03.009. Epub 2020 Apr 15. No abstract available. PMID 32305473
- [Background] Arbelo E, Protonotarios A, Gimeno JR, Arbustini E, Barriales-Villa R, Basso C, Bezzina CR, Biagini E, Blom NA, de Boer RA, De Winter T, Elliott PM, Flather M, Garcia-Pavia P, Haugaa KH, Ingles J, Jurcut RO, Klaassen S, Limongelli G, Loeys B, Mogensen J, Olivotto I, Pantazis A, Sharma S, Van Tintelen JP, Ware JS, Kaski JP; ESC Scientific Document Group. 2023 ESC Guidelines for the management of cardiomyopathies. Eur Heart J. 2023 Oct 1;44(37):3503-3626. doi: 10.1093/eurheartj/ehad194. No abstract available. PMID 37622657
- [Background] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Granger CB, Hammill SC, Hlatky MA, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS Guideline for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2018 Oct 2;72(14):e91-e220. doi: 10.1016/j.jacc.2017.10.054. Epub 2018 Aug 16. No abstract available. PMID 29097296
- [Background] Frustaci A, Russo MA, Chimenti C. Randomized study on the efficacy of immunosuppressive therapy in patients with virus-negative inflammatory cardiomyopathy: the TIMIC study. Eur Heart J. 2009 Aug;30(16):1995-2002. doi: 10.1093/eurheartj/ehp249. Epub 2009 Jun 25. PMID 19556262
- [Background] Chimenti C, Russo MA, Frustaci A. Immunosuppressive therapy in virus-negative inflammatory cardiomyopathy: 20-year follow-up of the TIMIC trial. Eur Heart J. 2022 Sep 21;43(36):3463-3473. doi: 10.1093/eurheartj/ehac348. PMID 35831932
- [Background] Koplan BA, Soejima K, Baughman K, Epstein LM, Stevenson WG. Refractory ventricular tachycardia secondary to cardiac sarcoid: electrophysiologic characteristics, mapping, and ablation. Heart Rhythm. 2006 Aug;3(8):924-9. doi: 10.1016/j.hrthm.2006.03.031. Epub 2006 Mar 30. PMID 16876741
- [Background] Uusimaa P, Ylitalo K, Anttonen O, Kerola T, Virtanen V, Paakko E, Raatikainen P. Ventricular tachyarrhythmia as a primary presentation of sarcoidosis. Europace. 2008 Jun;10(6):760-6. doi: 10.1093/europace/eun110. Epub 2008 May 2. PMID 18456644
- [Background] Peretto G, Sala S, Rizzo S, De Luca G, Campochiaro C, Sartorelli S, Benedetti G, Palmisano A, Esposito A, Tresoldi M, Thiene G, Basso C, Della Bella P. Arrhythmias in myocarditis: State of the art. Heart Rhythm. 2019 May;16(5):793-801. doi: 10.1016/j.hrthm.2018.11.024. Epub 2018 Nov 24. PMID 30476544